CLINICAL TRIAL: NCT01943344
Title: Safety and Performance Study of Large Hole Vascular Closure Device - FRONTIER I Study
Brief Title: Safety and Performance Study of Large Hole Vascular Closure Device
Acronym: FRONTIER-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivasure Medical Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P043-00; EUDAMED: CIV-IE-13-01-009581 (Other: Irish Medicines Board)
Record Dates: First submitted 2013-09-11; First posted 2013-09-16 (Estimated); Results first posted 2016-07-06 (Estimated); Last update posted 2018-11-02 (Actual); Status verified 2018-01

CONDITIONS: Percutaneous Closure of Arteriotomy in Common Femoral Artery
Keywords: vascular large hole closure; arteriotomy closure; Large hole vascular closure device; vascular closure device; percutaneous vascular closure device

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (Experimental): Subjects that receive VIVASURE CLOSURE DEVICE™
  Interventions: Device: VIVASURE CLOSURE DEVICE™

INTERVENTIONS:
Device: VIVASURE CLOSURE DEVICE™ — implantation of VIVASURE CLOSURE DEVICE™
  Other Names: DP2; DP2-FA1-1

SUMMARY:
The purpose of this Clinical Investigation is to gather feasibility data on the clinical use of the VIVASURE CLOSURE DEVICE™ in relation to safety, and to confirm its performance to percutaneously close femoral arterial puncture sites in the range of 18-24 F, post endovascular procedures.

DETAILED DESCRIPTION:
This study will be a prospective, multi-centred, non-randomized pilot study to investigate the safety and performance of the VIVASURE CLOSURE DEVICE™. All patients undergoing a procedure requiring an arteriotomy in the range of 18 to 24 F, via the common femoral artery will be screened against the inclusion/exclusion criteria. If the patient meets the requirements of the clinical investigation, they shall be invited to participate, provide informed consent and shall subsequently be assigned a subject number.

Patient safety will be monitored closely by the Data Safety Monitoring Committee (DSMC). Safety data will be reported to the DSMC for every patient with a reported complication. The DSMC will adjudicate on the safety data to determine whether it is safe to continue enrolment.

Subjects shall have a 1, 3 and 12 month follow-up assessment. Safety data from the follow-ups will be assessed by the Data Safety Monitoring Committee.

This protocol will adopt the VARC-2 definitions for major vascular complication associated with closure of the access site.

This pilot study will enrol approximately 10 subjects. The study is designed to support a larger CE Mark study. As such, a study safety assessment will be complete when all patients have completed their 1 month follow-up assessment. The Data Safety Monitoring Committee (DSMC) will review all complications and recommend whether it is safe to proceed to the CE Mark study. All patients will continue to be followed at 1, 3 and 12 month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age.
* Each patient, or his or her guardian or legal representative, is willing to give informed consent.
* Clinically indicated for an endovascular procedure involving access through the femoral artery, with an access puncture of 18 - 24 F.
* Females who are not pregnant or lactating, and not planning to become pregnant ≤ 12 months. A pregnancy test may be performed to confirm this.

Exclusion Criteria:

There will be no exclusion of patients from this trial in respect of race, co-existent disease or concomitant therapy, with the exception of those listed below.

* Severe acute non-cardiac systemic disease or terminal illness with a life expectancy of less than one year.
* Evidence of systemic bacterial or cutaneous infection, including groin infection.
* Evidence of MRSA (Methicillin-resistant Staphylococcus aureus) and/or VRE (vancomycin-resistant Enterococci) colonisation.
* With arterial access other than the common femoral artery.*
* Patients suffering with definitive or potential coagulopathy or platelet count less than 100,000/µl.
* Patient with a haematocrit of less than 32 %.
* A measured activated clotting time (ACT) of greater than 350 seconds immediately prior to sheath removal.*
* If patients are expected to be continuously treated with anticoagulation therapy post-procedure such that their ACT reading is expected to be elevated above 350 seconds for more than 24 hours after the procedure.
* Evidence of arterial diameter stenosis greater than 20 % within 20 mm of the arteriotomy.*
* Circumferential calcification within 20 mm of the arteriotomy.*
* Use of systemic thrombolytic agents within 24 hours prior to or during the catheterisation procedure which cause the concentration of fibrinogen to be less than 100 mg/dl.
* Patients in which the arteriotomy is less than 18 F or greater than 24 F.*
* Known allergy to any of the materials used in the device (Refer to Instructions for Use).
* Currently enrolled in any other investigational clinical study, where the primary endpoint has not yet been achieved.
* Patients judged unsuitable for surgical repair of the access site.
* If puncture site is via a vascular graft.
* If there is any indication that the puncture has been made in the profunda femoris or located less than 10 mm above the profunda femoris.*
* Patients with a common femoral artery lumen diameter of less than 7 mm.
* Patients that have a lower extremity amputation from an access site limb.
* Patients that have undergone a percutaneous procedure using a non-absorbable vascular closure device (excluding suture mediated) for haemostasis in the ipsilateral leg.
* Patients that have undergone a percutaneous procedure greater than 8 F in the ipsilateral leg, within the previous 90 days.
* Patients that have undergone a percutaneous procedure of 8 F or less using an absorbable intravascular closure device for haemostasis, in the ipsilateral leg, within the previous 90 days.
* Patients that have undergone a percutaneous procedure of 8 F or less using a suture mediated closure device for haemostasis, in the ipsilateral leg, within the previous 30 days.
* Patients that have undergone a percutaneous procedure of 8 F or less using manual/mechanical pressure for haemostasis in the ipsilateral leg, within the previous 30 days.
* Patients with an acute haematoma of any size, arteriovenous fistula or Pseudoaneurysm at the access site.*
* Significant blood loss/transfusion during interventional procedure or within 20 days prior to procedure requiring transfusion of greater than 4 units of blood.*
* Angiographic evidence of arterial laceration, dissection or stenosis within the external iliac or femoral artery before the use of the VCD.*

  * May not be known until after the patient has given informed consent and the procedure has started.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-07; Primary Completion 2014-07 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Peter Crean, FRCPI MB ChB, Principal Investigator — St Jame's Hospital, Dublin
Locations (1):
- St Jame's Hospital, Dublin, Ireland

RESULTS

PARTICIPANT FLOW:
Groups:
- Closure Device: Subjects that receive VIVASURE CLOSURE DEVICE™
  VIVASURE CLOSURE DEVICE™: implantation of VIVASURE CLOSURE DEVICE™
Period: Overall Study
Arm/Group | Closure Device
Started | 12
Completed | 9
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 12
Age, Continuous [Mean (Full Range); unit: years] | 78 [66 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 9
Region of Enrollment [Number; unit: participants]
  Ireland | 12

OUTCOME MEASURES:

1. Primary Outcome: Major Vascular Complications Directly Related to Device
Description: Major complication rates directly related to the VIVASURE CLOSURE DEVICE™ up to 3 months from implantation, (as defined by VARC-2).
Time Frame: up to 3 Months of implantation
Population: Two subjects died prior to 3-month follow-up, not related to the study device, hence, were not included in analysis. A third subject died prior to study completion (12 month follow-up), not related to the study device.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment
Number analyzed (Participants) | 10
percentage of participants | 0

2. Secondary Outcome: Minor Vascular Complications Directly Related to Device
Description: Incidence of minor complications directly related to the VIVASURE CLOSURE DEVICE™ up to 3 months from implantation, as defined by VARC-2.
Time Frame: up to 3 months from implantation
Population: as for outcome 1
Measure: Number; unit: percentage of Participants
Groups:
- Teatment: Subjects that receive VIVASURE CLOSURE DEVICE™
  VIVASURE CLOSURE DEVICE™: implantation of VIVASURE CLOSURE DEVICE™
Arm/Group | Teatment
Number analyzed (Participants) | 10
percentage of Participants | 0

3. Other Pre Specified Outcome: Performance
Description: Assessed by technical success rate for the VIVASURE CLOSURE DEVICE™ (Tech Success: haemostasis by investigational device, not leading to alternative treatment other than manual compression or adjunctive endovascular ballooning)
Time Frame: up to 3 month of implantation
Population: All subjects entered into study that received the Vivasure Closure Device or had intension to treat with the Vivasure Closure Device.
Measure: Number; unit: percentage of successful deployments
Arm/Group | Treatment
Number analyzed (Participants) | 12
percentage of successful deployments | 100

ADVERSE EVENTS:
Arm/Group | Treatment
Serious Adverse Events (participants affected / at risk) | 6/12
Other Adverse Events (participants affected / at risk) | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=12)
Cardiac tamponade (Cardiac disorders) | 1 (1) — Not related to study device
Cardiogenic shock (Cardiac disorders) | 1 (1) — Not related to study device
COPD (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to study device
Chronic heart failure (Cardiac disorders) | 4 (6) — Not related to study device
Septicemia/bacteremia (Infections and infestations) | 1 (1) — Not related to study device
Renal failure/insufficency (Renal and urinary disorders) | 1 (1) — Not related to study device
Lower respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to study device
Anemia (Blood and lymphatic system disorders) | 1 (1) — Not related to study device
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Not related to study device
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not related to study device

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No